CLINICAL TRIAL: NCT04592172
Title: Impact of Bedtime Routines on Sleep and Development in Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Joseph's University, Philadelphia (Other)
Collaborators: Temple University (Other); Simms/Mann Family Foundation (Unknown); CuddleBright Cares (Unknown); Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02
Record Dates: First submitted 2020-09-04; First posted 2020-10-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Sleep Disturbance; Child Development
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: 100 caregiver-infant dyads (infants ages 12.0 to 14.9 months) will be recruited from Temple Pediatric Care Outpatient Pediatric office with follow-up visits at approximately 15 and 24 months of age.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bedtime Routine Education (Experimental): 50 families will be randomly assigned to receive the bedtime routine intervention, 3 Cs for Bedtime ZZZs delivered by research assistants at the 12-month and 15-month well-child visits, in additional to receiving usual clinical care. The intervention will take approximately 30-45 minutes to implement at each study visit. Research assistants will be trained and supervised by board-certified Behavioral Sleep Medicine providers. This intervention focuses on developing an individualized bedtime routine, including such activities as a bath, teeth-brushing, reading stories, singing songs, and cuddling, based on parent's preferences. Families will receive appropriate materials for their bedtime routine, including a CuddleBright kit, bedtime books, toothbrush/toothpaste, and the created bedtime chart to take home.
  Interventions: Behavioral: Bedtime Routine Education
- Control group (No Intervention): 50 families will be randomly assigned to control group (usual care).

INTERVENTIONS:
Behavioral: Bedtime Routine Education — The intervention aims to promote healthy sleep and improved developmental outcomes in infants. Individualized bedtime routine education, including such activities as a bath, teeth-brushing, reading stories, singing songs, and cuddling will be implemented by research assistants at the 12-month well-child visit. Reinforcement of the bedtime routine education will be implemented at the 15-month visit. Each individualized bedtime routine will incorporate 3-5 steps and a bedtime routine chart depicting those steps will be created and provided to the families. Families will receive materials for their bedtime routines, including a CuddleBright kit, 1-2 additional bedtime books, toothbrush/toothpaste , and the created bedtime chart. On top of that, families will also receive a children's book provided by Reach Out and Read through the study period.
  Arms: Bedtime Routine Education

SUMMARY:
Investigators will recruit up to 100 families (children aged 12.0 to 14.9 months and their primary caregivers) at their scheduled 12-month well child care infant visit at Temple Pediatric Care. The purpose of this randomized controlled trial is to examine the impact of implementation of a bedtime routine program, Connect, Calm, & Comfort: 3 Cs for Bedtime ZZZs, to promote better sleep and improve developmental outcomes in toddlers from primarily low-income families.

DETAILED DESCRIPTION:
A bedtime routine is a key factor in the promotion of not only healthy sleep, but also potentially of broad development and wellbeing in early childhood. A bedtime routine, in and of itself, embodies the characteristics of nurturing care and early child stimulation especially for at-risk children. It is consistent with the Lancet Early Childhood Series Steering Committee emphasizing the need for nurturing care, which includes adequate health, nutrition, security and safety, responsive caregiving, and early learning opportunities, to help young children (ages 0-5 years) reach their full developmental potential, and to build a strong foundation for subsequent development, health, and wellbeing. Common, adaptive components of a bedtime routine can contribute to an array of positive developmental outcomes beyond improved sleep, inclusive of language development, literacy, child emotional and behavioral regulation, parent-child attachment, and family functioning, among other outcomes. Although studies have been conducted on the relationship between bedtime routines and sleep, there have been few studies looking at bedtime routines and other developmental outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to a well child visit
* Child between 12.0 to 14.9 months of age
* English-speaking
* Caregiver is legal guardian of infant
* Caregiver is primary caregiver of infant

Exclusion Criteria:

* Non-English speaking
* Absence of primary caregiver at both the 12-month and 15-month well-child visit

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Change in sleep outcomes - bedtime routines | 12-month, 15-month, and 24-month visits
  At the 12-month, 15-month, and 24-month visits, caregivers will report on bedtime routine frequency (the number of nights their child followed the same bedtime routine) from the well-validated and widely used Brief Infant Sleep Questionnaire-Revised (Short Form) (BISQ-R).
Sleep outcomes - patterns and problems | 15-month and 24-month visits
  At 15-month and 24-month visits, caregivers will complete the well-validated and widely used Brief Infant Sleep Questionnaire-Revised (Short Form) (BISQ-R) to report on toddler sleep over the last two weeks. The BISQ-R contains items related to the child sleep environment (e.g., sleep space, location, and arrangement) and patterns (e.g., bedtime, sleep onset latency, night awakening frequency and duration, wake time). Items also assess caregiver-perceived child sleep problems (e.g., overall sleep problem severity, bedtime resistance severity).

SECONDARY OUTCOMES:
Socio-emotional outcomes | 15-month and 24-month visits
  The Brief Infant-Toddler Social and Emotional Assessment (BITSEA) is a screener derived from the longer ITSEA. It is a parent questionnaire that assesses the social-emotional development of children ranging in age from 12 to 36 months. Caregivers will rate each statement that best describes the child's behavior in the past month, with scores ranging from 0 to 84. Higher scores denote possible social-emotional/ behavioral concerns.
Parent stress | 15-month and 24-month visits
  The Parenting Stress Index (PSI) Short form is a 36-items reliable measure to assess total parenting stress with high internal consistency. It consists of three subscales: parental distress, parent-child dysfunctional interaction, and difficult child. Statements on this measure are rated on a 5-point Likert scale from strongly agree to strongly disagree, with scores ranging from 36 to 180. Higher scores denote higher level of stress in parent-child relationship.
Treatment acceptability | 15-month and 24-month visits
  Caregivers randomized to the bedtime routine education arm will complete the treatment acceptability/bedtime routine evaluation form. Caregivers will rate 7 statements related to the perceived helpfulness/efficacy and acceptability of the intervention using a 5-point Likert scale from strongly disagree to strongly agree, with total scores ranging from 0 to 35. Higher scores indicate higher perceived helpfulness and acceptability of the intervention.
Treatment feasibility | 12-month and 15-month visits
  The study team will track the number of treatment sessions completed (maximum = 2, 1 session at 12-month visit and 1 session at 15-month visit) for caregivers randomized to the bedtime routine education arm.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Heere, MD, Principal Investigator — Temple University
Locations (1):
- Temple Pediatrics, Philadelphia, Pennsylvania, United States